CLINICAL TRIAL: NCT06358183
Title: Comprehensive Analysis of Emergency and Essential Surgical Capacity in Zimbabwean Public Hospitals: A National Cross-sectional Survey
Brief Title: Surgical Capacity in Zimbabwean Public Hospitals
Status: Completed | Type: Observational
Sponsor: Parirenyatwa Hospital (Other)
Responsible Party: Principal Investigator, Dennis Mazingi, Hospital Medical Officer, Parirenyatwa Hospital
Other Study IDs: ESC001
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Surgery; Anesthesia
Keywords: Global surgery; Surgical capacity; Zimbabwe

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — no intervention used

SUMMARY:
This study aimed to understand how ready Zimbabwe's public hospitals are to perform essential surgeries, which are critical for treating a wide range of health issues from emergencies like car accidents to planned procedures such as childbirth by caesarean section. The researchers looked at hospitals across Zimbabwe to see what kind of surgery facilities, equipment, and specialists were available.

DETAILED DESCRIPTION:
Abstract Background: Access to surgical care is an essential component of universal health coverage, but surgical capacity is lacking in many low- and middle-income countries. Surgical capacity in Zimbabwe, a lower-middle income country, is undocumented. The objective of this study was to assess surgical capacity in public hospitals in Zimbabwe.

Methods: A national hospital survey was performed in 2019 using a validated surgical situational analysis tool. the investigators included district, provincial and central hospitals in the public sector across all 10 provinces of Zimbabwe. Data was collected from key informants using an online survey. information gathered included an inventory of infrastructural components required to perform essential surgical services, a survey of healthcare workers involved in surgical care (the Surgical Anaesthetic and Obstetric workforce); a submission of the number of surgical procedures including bellwether procedures performed over the course of the last year and also surgical sundries and consumables required to perform surgical services.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals were considered eligible if there was any major or minor surgical activity occurring in the facility

Exclusion Criteria:

* hospitals dedicated to a non-surgical pursuit
* private hospitals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: public hospitals in zimbabwe
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Bellwether procedures | in 1 calendar year
  number of bellwether procedures performed in each hospital
Procedures | in 1 calendar year
  number of other procedures performed in each hospital
SAO density | in 1 calendar year
  Number of surgical anesthetic and obstetric practitioners per 100 000 population
Infrastructure | in 1 calendar year
  Availability of basic and specific infrastructure in each hospital

CONTACTS AND LOCATIONS:
Overall Officials: Shingai Nyaguse-Chiurunge, Study Director — Parirenyatwa
Locations (1):
- Parirenyatwa Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No